CLINICAL TRIAL: NCT04765241
Title: Adolescents and Young Adults Becoming Physically Active After Cancer Trial
Brief Title: mHealth Physical Activity Intervention for Young Cancer Survivors
Acronym: AYA-PACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HREBA.CC-20-0397
Record Dates: First submitted 2021-02-09; First posted 2021-02-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Adolescent cancer; Young adult cancer; Physical activity; mHealth; Survivorship; AYA cancer
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study team, with the exception of the study coordinator, will be blinded to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Physical Activity Intervention (Experimental): The intervention arm will receive a 12 month mobile health (mHealth) physical activity intervention with a goal of increasing their moderate-vigorous intensity physical activity levels by 90 minutes per week above baseline
  Interventions: Behavioral: Physical Activity
- Control (No Intervention): Controls will receive general health education materials

INTERVENTIONS:
Behavioral: Physical Activity — The intervention includes a physical activity prescription, a Polar activity tracker watch, access to a private AYA cancer survivor community through the Polar Flow community platform, mHealth nudges and surveys via text messaging, and regular phone or email contact from study staff.
  Arms: mHealth Physical Activity Intervention

SUMMARY:
In this randomized controlled trial the investigators will determine whether a mobile health intervention can increase physical activity levels in AYA cancer survivors over a one year period. The investigators will recruit 320 cancer survivors in Alberta who were diagnosed with a first cancer between the ages of 15 to 39 years and are within one year of treatment completion. Participants will be randomized into either the control group (educational information) or the intervention group (educational information; personalized physical activity plan; activity tracker watch; access to a private, online survivor community; motivational text messages and check-in calls/e-mails). All participants will complete fitness testing and questionnaires at baseline, 6 months and 12 months. A final measurement at 24 months will test long-term effectiveness.

DETAILED DESCRIPTION:
Background:

There is a need for adolescent and young adult (AYA) cancer research because the number of new cancers in young people is increasing and the survivor population is growing. Interventions that try to reduce problems that affect people after cancer are particularly important since its treatments can have negative effects on survivors' physical and mental health even decades after diagnosis.

Aim:

Given the many positive effects of physical activity (e.g. improved fitness and quality of life), the study aims to encourage AYA cancer survivors to be more physically active as they shift from treatment to survivorship care. The main goal of this study is to see if a home-based, mobile health (mHealth) physical activity intervention can increase physical activity levels by at least 90 minutes/week compared to baseline in AYA cancer survivors.

Methods:

The investigators will conduct a two-center randomized controlled trial of 320 AYA cancer survivors. Participants (N=320) will be Albertan residents, diagnosed with a first cancer between the ages of 15 and 39 years, and within one year of cancer treatment completion. At the start of the study, participants will complete fitness testing and questionnaires. Participants will then be randomly put into either a control or intervention group. The control group will receive educational information only. The intervention group will also receive a personalized physical activity plan, an activity tracker watch, access to a private, online survivor community, motivational text messages and check-in calls/e-mails. Fitness testing and questionnaires will be repeated at 6 and 12 months to see if the intervention increased physical activity levels and improved health outcomes among the participants in the intervention group compared to controls. A final measurement at 24 months will test long-term use.

ELIGIBILITY:
Inclusion Criteria:

* Lives in Alberta
* Diagnosed with invasive malignancy in Alberta
* Completed active cancer directed therapy (cytotoxic chemotherapy, radiation therapy and/or definitive surgical intervention) in the last 12 months, except for "maintenance" therapy to prevent recurrences
* Have the ability to read, write and speak English
* Have access to the Internet on at least a weekly basis
* Have a mobile phone with a text messaging plan
* Willing to be randomized to either arm.

Exclusion Criteria:

* Health problems which preclude the ability to walk for physical activity, as measured by the Physical Activity Readiness Questionnaire (PAR-Q)
* Currently pregnant or planning to become pregnant within the next 6 months
* Currently taking part in > 300 minutes/week of moderate-to-vigorous intensity physical activity on a regular basis

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 287 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in weekly minutes of moderate-vigorous intensity physical activity | Baseline, 6 months, 12 months, 24 months
  Measured by Actigraph

SECONDARY OUTCOMES:
Changes in weekly minutes of sedentary time | Baseline, 6 months,12 months
  Measured by Actigraph
Changes in weekly minutes of sleep | Baseline, 6 months,12 months
  Measured by Actigraph
Changes in the Pittsburgh Sleep Quality Index (PSQI) Global Sleep Quality Score | Baseline, 6 months,12 months
  Global score range is 0 to 23 where higher scores indicate worse sleep quality
Changes in weight | Baseline, 6 months,12 months
  Measured in kilograms
Changes in body mass index (BMI) | Baseline, 6 months,12 months
  Measured by combining height (meters) and weight (kilograms) and reported in kg/m2
Changes in waist and hip circumference | Baseline, 6 months,12 months
  Measured in centimeters
Changes in cardiorespiratory fitness | Baseline, 6 months,12 months
  Measured by peak oxygen consumption in relative (ml/kg/min) values using the incremental Balke and Ware treadmill test with direct measures of gas exchange and ventilation
Changes in cardiorespiratory fitness | Baseline, 6 months,12 months
  Measured by peak oxygen consumption in absolute (L/min) values using the incremental Balke and Ware treadmill test with direct measures of gas exchange and ventilation
Changes in grip strength | Baseline, 6 months,12 months
  Measured in kilograms using a hand dynamometer
Changes in upper body muscular strength | Baseline, 6 months,12 months
  Measured in kilograms using an 8-10 repetition maximum (RM) chest press test used to predict 1-RM
Changes in upper body muscular endurance | Baseline, 6 months,12 months
  Measured in kilograms using the maximum number of chest press repetitions completed at 50-70% of estimated 1-RM
Changes in lower body muscular strength | Baseline, 6 months,12 months
  Measured in kilograms using an 8-10 repetition maximum (RM) leg press test used to predict 1-RM
Changes in lower body muscular endurance | Baseline, 6 months,12 months
  Measured in kilograms using the maximum number of leg press repetitions completed at 50-70% of estimated 1-RM
Changes in frailty | Baseline, 6 months,12 months
  Defined according to the Fried phenotype which takes into account low lean muscle mass, exhaustion, low energy expenditure, walking limitations, and weakness
Changes in the Short Form 36 (SF-36) Mental Health Component subscale | Baseline, 6 months,12 months
  Score range is from 0 to 100 where higher scores indicate better mental health
Changes in the Short Form 36 (SF-36) Physical Health Component subscale | Baseline, 6 months,12 months
  Score range is from 0 to 100 where higher scores indicate better physical health
Changes in the Short Form 36 (SF-36) Physical Functioning subscale | Baseline, 6 months,12 months
  Score range is from 0 to 100 where higher scores indicate higher functioning
Changes in the Short Form 36 (SF-36) Role-physical subscale | Baseline, 6 months,12 months
  Score range is from 0 to 100 where higher scores indicate higher functioning
Changes in the Short Form 36 (SF-36) Bodily Pain subscale | Baseline, 6 months,12 months
  Score range is from 0 to 100 where higher scores indicate less pain
Changes in the Short Form 36 (SF-36) General Health subscale | Baseline, 6 months,12 months
  Score range is from 0 to 100 where higher scores indicate better health
Changes in the Short Form 36 (SF-36) Vitality subscale | Baseline, 6 months,12 months
  Score range is from 0 to 100 where higher scores indicate higher vitality
Changes in the Short Form 36 (SF-36) Social Functioning subscale | Baseline, 6 months,12 months
  Score range is from 0 to 100 where higher scores indicate higher functioning
Changes in the Short Form 36 (SF-36) Role-emotional subscale | Baseline, 6 months,12 months
  Score range is from 0 to 100 where higher scores indicate higher functioning
Changes in the Short Form 36 Mental Health subscale | Baseline, 6 months,12 months
  Score range is from 0 to 100 where higher scores indicate better mental health
Changes in the Cancer Distress Scales for AYAs Impact of Cancer subscale | Baseline, 6 months,12 months
  Scores range from 0 to 100 where higher scores indicate more distress
Changes in the Cancer Distress Scales for AYAs Physical subscale | Baseline, 6 months,12 months
  Scores range from 0 to 100 where higher scores indicate more distress
Changes in the Cancer Distress Scales for AYAs Emotional subscale | Baseline, 6 months,12 months
  Scores range from 0 to 100 where higher scores indicate more distress
Changes in the Cancer Distress Scales for AYAs Cognitive subscale | Baseline, 6 months,12 months
  Scores range from 0 to 100 where higher scores indicate more distress
Changes in the Cancer Distress Scales for AYAs Cancer Worry subscale | Baseline, 6 months,12 months
  Scores range from 0 to 100 where higher scores indicate more distress
Changes in the Cancer Distress Scales for AYAs Employment subscale | Baseline, 6 months,12 months
  Scores range from 0 to 100 where higher scores indicate more distress
Changes in the Cancer Distress Scales for AYAs Education subscale | Baseline, 6 months,12 months
  Scores range from 0 to 100 where higher scores indicate more distress
Changes in the Cancer Distress Scales for AYAs Practical subscale | Baseline, 6 months,12 months
  Scores range from 0 to 100 where higher scores indicate more distress
Changes in the Functional Assessment of Cancer Therapy Cognitive Function Perceived Cognitive Impairment subscale | Baseline, 6 months,12 months
  Score range is from 0 to 80. Higher scores indicate poorer quality of life.
Changes in the Functional Assessment of Cancer Therapy Cognitive Function (FACT-Cog) Comments From Others subscale | Baseline, 6 months,12 months
  Score range is from 0 to 16 where higher scores indicate poorer cognition
Changes in the Functional Assessment of Cancer Therapy Cognitive Function (FACT-Cog) Perceived Cognitive Abilities subscale | Baseline, 6 months,12 months
  Score range is from 0 to 36 where higher scores indicate poorer cognition
Changes in the Functional Assessment of Cancer Therapy Cognitive Function (FACT-Cog) Impact on Quality of Life subscale | Baseline, 6 months,12 months
  Score range is from 0 to 16 where higher scores indicate poorer cognition
Changes in the Functional Assessment of Cancer Therapy Fatigue (FACT-F) | Baseline, 6 months,12 months
  Score range is from 0 to 52 where higher scores indicate less fatigue
Changes in the Comprehensive Score for Financial Toxicity (COST) | Baseline, 6 months,12 months
  Score range is from 0 to 44 where higher scores indicate better financial wellbeing

CONTACTS AND LOCATIONS:
Overall Officials: Christine Friedenreich, Study Director — Cancer Care Alberta; Miranda Fidler-Benaoudia, Principal Investigator — Cancer Care Alberta
Locations (1):
- Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No